CLINICAL TRIAL: NCT05236556
Title: Supporting Use of AC Through Provider Profiling of Oral AC Therapy for AF IV
Acronym: SUPPORT-AF IV
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: University of Florida (Other)
Responsible Party: Principal Investigator, Alok Kapoor, Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HL155343
Record Dates: First submitted 2022-02-01; First posted 2022-02-11 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: After removing providers who opted out, the investigators will randomize the remaining providers to either intervention or control in a 1:1 ratio, using randomly permuted blocks; randomization will be stratified jointly by provider type (cardiologist/primary care provider) and study site (University of Massachusetts/University of Florida). The allocation of the provider conducting the first visit for a patient will dictate the allocation for the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Receive best practice advisory (BPA)
  Interventions: Behavioral: Best practice advisory (BPA)
- Control (No Intervention): Does not receive best practice advisory (BPA)

INTERVENTIONS:
Behavioral: Best practice advisory (BPA) — For patients who are not on oral anticoagulation (AC) but have elevated stroke risk, the practice advisory will "fire," which is to say it will be active in the providers workflow during outpatient encounters with a patient's primary care provider (PCP) or cardiology provider.
  Arms: Intervention

SUMMARY:
Six million Americans live with atrial fibrillation (AF), a heart rhythm abnormality that is a major risk factor for stroke and only half of those AF patients receive oral anticoagulation (AC). Within the context of an ongoing collaboration between two large learning health systems, the investigators propose to study the impact of a shared clinical decision support tool embedded within the electronic health record designed to enhance guideline-based AC prescription. The hypothesis the investigators are testing is that the number of AC starts in patients seen by intervention providers will be higher than in patients seen by control providers. Additionally, the investigators are testing the hypothesis that the risk of not persisting on AC will be higher in the patients of control providers compared with patients of intervention providers.

DETAILED DESCRIPTION:
The proposed project will examine the impact of a novel anticoagulant (AC) clinical decision support tool within the electronic health record (EHR) on AC prescribing behaviors among healthcare providers from two distinct health systems who receive it. Using a mixed-methods approach, the investigators will also examine how healthcare providers interact with the decision support tool to further refine the tool and measure its impact on anticoagulation prescribing behaviors. The investigators will also examine clinician engagement through provider interviews and detailed study of behaviors using electronic health record access logs. Finally, the investigators will refine the alert, develop a comprehensive dissemination plan, and create an implementation toolkit to widen the use of the alert at other learning health systems nationally.

After identifying a list of all cardiology providers and primary care providers (PCPs), the investigators will send an email to all providers notifying them of our research study and request for participation. The investigators will send this email through our data collection platform- Redcap-with a link to one item survey allowing providers to opt out. This follows the prior SUPPORT-AF II protocol which the investigators' Institutional Review Board (IRB) approved. Based on discussions with the IRB, the investigators do not anticipate requiring informed consent from providers or patients for executing this aim of the proposal. After removing providers who opted out, the investigators will randomize the remaining providers to either intervention or control in a 1:1 ratio, using randomly permuted blocks; randomization will be stratified jointly by provider type (cardiologist / PCP) and study site (University of Massachusetts/University of Florida). The allocation of the provider conducting the first visit for a patient will dictate the allocation for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Providers caring for patients aged 18 years and older with international classification of disease 10th revision (ICD-10) diagnostic code consistent with atrial fibrillation (AF) or atrial flutter who had a visit with a primary care provider or cardiovascular medicine specialist in the previous one year with the diagnosis of AF present as an active diagnosis in the electronic health record (EHR).
* Patients aged 18 years and older with ICD-10 diagnostic code consistent with AF or atrial flutter who had a visit with a primary care provider or cardiovascular medicine specialist in the previous one year with the diagnosis of AF present as an active diagnosis in the EHR.

Exclusion Criteria:

* Left atrial appendage closure
* Hospice status
* Providers who do not care for patients aged 18 years and older with ICD-10 diagnostic code consistent with AF or atrial flutter who had a visit with a primary care provider or cardiovascular medicine specialist in the previous one year with the diagnosis of AF present as an active diagnosis in the EHR.
* Patients under the age of 18; patients without a ICD-10 diagnostic code consistent with AF or atrial flutter who had a visit with a primary care provider or cardiovascular medicine specialist in the previous one year with the diagnosis of AF present as an active diagnosis in the EHR. Patients will also be excluded from this study if they are known to be pregnant or a prisoner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5094 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Initiation of Oral Anticoagulation (AC) Use | 12 months
  The number of participants who initiate AC will be measured using the first encounter for each participant in the 12 months after randomization of providers and launch of the enhanced alert. To count as an AC initiation, a participant will have to have presence of an anticoagulant on his/her current medication list or an international normalized ratio (INR) lab value 1.5 or greater in the two months following the index encounter.
Length of Duration for Oral Anticoagulation (AC) Use | 12 months
  The number of days participants continue on AC for one year after AC initiation will be tracked. Up to one month off AC such as for bleeding or surgical procedure will be permitted so long as the participant resumes AC prior to the end of the 12 month follow up.

SECONDARY OUTCOMES:
Hospitalization for new Stroke, Transient Ischemic Attack, or Systemic Embolism Ischemic Attack /Systemic Embolism. | 12 months
  The number of new hospitalizations for participants for strokes, transient ischemic attacks, or systemic embolisms that is determined by international classification of disease (ICD) codes in the medical record. The count of new hospitalizations for strokes will be limited to those hospitalizations with the stroke code as the admitting or principal diagnosis code. Verification will be performed through manual chart review.
Incidence of Major Hemorrhage and Clinically Relevant non-major Bleeding | 12 months
  Bleeding events will be quantified using international classification of disease (ICD) codes if a bleeding code is present in the admitting or principal diagnosis fields. Verification will be performed through manual chart review.

CONTACTS AND LOCATIONS:
Overall Officials: Alok Kapoor, MD, Principal Investigator — UMass Chan Medical School
Locations (2):
- United States (2):
  - University of Florida College of Medicine - Jacksonville, Jacksonville, Florida
  - UMass Chan Medical School, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: No